CLINICAL TRIAL: NCT01972191
Title: Comparison of Three Corneal Horizontal Marking Techniques Using iTrace™
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2013-0049
Record Dates: First submitted 2013-10-15; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Corneal Horizontal Marking.
Keywords: Toric marking, Corneal horizontal marking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Group 1 : Bare eye marking group
- Group 2: Group 2 : Pendulum attached marker group
- Group 3: Group 3 : Horizontal slit beam assisted marker group

SUMMARY:
Before astigmatism reducing surgery, accurate corneal horizontal marking before surgery is important. Due to new corneal topographic method, iTrace™ surgical workstation, precise evaluation of corneal horizontal marking is available. In this study the investigators compared three known corneal horizontal making techniques and evaluate accuracy of each methods using iTrace™.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled to have cataract surgery
* Age between 50 to 85 years

Exclusion Criteria:

* With an underlying corneal or conjunctival disorder

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Who visited professor Tae Im Kim's clinic, department of ophthalmology, Severance hospital.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The vertical height deviation and rotational axis misalignment amount of each three marking techniques, evaluated by iTrace surgical workstation. | Within 10 minutes after corneal horizontal marking.
  Nasal and temporal marked spots saved in iTrace surgical workstation program.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Hoffer KJ. Biometry of 7,500 cataractous eyes. Am J Ophthalmol. 1980 Sep;90(3):360-8. doi: 10.1016/s0002-9394(14)74917-7. No abstract available. PMID 7425052
- [Background] Cha D, Kang SY, Kim SH, Song JS, Kim HM. New axis-marking method for a toric intraocular lens: mapping method. J Refract Surg. 2011 May;27(5):375-9. doi: 10.3928/1081597X-20101005-01. Epub 2010 Oct 15. PMID 20954592